CLINICAL TRIAL: NCT02806154
Title: Frailty and Body Composition in the Elderly Cancer Patients Treated With Chemotherapy
Acronym: FRACTION
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/15/7831
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Cancer
Keywords: Cancer; Chemotherapy toxicity; Elderly patients; DEXA; muscle mass
MeSH Terms: conditions — Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly cancer patients: Elderly cancer patients treated with chemotherapy will have DEXA
  Interventions: Other: DEXA

INTERVENTIONS:
Other: DEXA — The appendicular muscle mass measured by DEXA
  Other Names: Dual Energy X-ray Absorptiometry

SUMMARY:
The investigators could hypothesize that age-related changes in body composition parameters play a role in the variable tolerance to chemotherapy in the elderly.

DETAILED DESCRIPTION:
However none of the studies relating body composition and chemotoxicity included elderly as a specific subpopulation. Furthermore in the majority of studies, body composition analyses are based on the estimation of muscle mass by CT scanner (axial L3 section). This method is to date not validated in the elderly cancer patients. Nevertheless some studies used Dual Energy X-ray Absorptiometry (DEXA), which is considered the gold standard in the assessment of body composition in older adults.

The investigators main hypothesis is that the appendicular muscle mass (I.e. muscle mass of the 4 limbs) operationalized as an index by dividing the muscle mass by squared height following Baumgartners' approach (Baumgartner, 1998) measured by DEXA (total of muscle mass of 4 limbs / height ²) represents a predictive factor of chemotoxicity in the elderly.

The finding that body composition is associated with poor tolerance of chemotherapy could lead to consider these parameters in the treatment decision of the elderly cancer patients and improve the current decision-making algorithms when treating older adults.

ELIGIBILITY:
Inclusion Criteria:

* Breast, prostate, bladder, colo-rectal, ovarian cancers, and lymphoma
* Metastatic or locally advanced neoplasm
* Initiation of first line chemotherapy
* Performance status World Health Organization (WHO) 0-3
* Capacity to give a written informed consent
* Life expectancy > 3 mouths

Exclusion Criteria:

* Concomitant targeted therapy
* Concomitant targeted radiotherapy
* Height > 196 cm, weight > 136 kg (DEXA not feasible)
* Hemopathy excluding lymphoma
* Cognitive impairment compromising the well proceeding and security of the study
* Cognitive impairment compromising the obtaining of a written informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly cancer patients treated with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by National Cancer Institute's - Common Toxicity Criteria (NCI-CTC) v4.0 | Up to 12 months
  Toxicity event defined by : first occurrence of grade 4 hematologic or grade 3-4 non hematologic toxicity as defined by the National Cancer Institute-Common Toxicity Criteria (NCI-CTC version 4) and/or disruption of chemotherapy because of inacceptable toxicity.

SECONDARY OUTCOMES:
Functional autonomy impairment | Up to 12 months
  defined as a loss of ≥ 0.5 point in Activities of Daily Living Scale.
Functional physical performances impairment | Up to 12 months
  defined as a loss ≥ 1 point in the Short Physical Performance Battery
Quality of life impairment | Up to 12 months
  defined as a loss ≥ 10 points in the EORTC quality of life questionnaire (QLQ) QLQ-C30 questionnaire
Early death | Up to 12 months
  defined by a death occuring during the 3 first months from the initiation of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Balardy, Principal Investigator — University Hospital, Toulouse
Locations (8):
- France (8):
  - Hôpital Sainte Marguerite, Marseille
  - CH de Montauban, Montauban
  - Institut du Cancer de Montpellier Val d'Aurelle, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital de Cimiez, CHU Nice, Nice
  - CH de Bigorre, Tarbes
  - Hospital of Toulouse, Toulouse
  - Institut Claudius Régaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinmeyer Z, Gerard S, Filleron T, Lozano S, Brechemier D, Abellan Van Kan G, Mourey L, Cristol-Dalstein L, De Decker L, Rolland Y, Balardy L. Low lean mass and chemotherapy toxicity risk in the elderly: the Fraction study protocol. BMC Cancer. 2019 Nov 27;19(1):1153. doi: 10.1186/s12885-019-6377-7. PMID 31775667